CLINICAL TRIAL: NCT01809028
Title: A Randomized Trial Evaluating the Number of Passes Required for Diagnostic Cell Block During Endoscopic Ultrasound-Fine Needle Aspiration of Solid Pancreatic Mass Lesions
Brief Title: Evaluating the Number of Passes Required for Diagnostic Cell Block During EUS-FNA of Solid Pancreatic Mass Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AdventHealth (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 407129
Record Dates: First submitted 2013-02-26; First posted 2013-03-12 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Pancreatic Cancer
Keywords: cell block, number of passes
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Endoscopic Ultrasound-Guided Fine Needle Aspiration; Biopsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EUS FNA with 2 passes (Active Comparator): biopsy with 2 passes of the needle
  Interventions: Procedure: EUS FNA with 2 passes
- EUS FNA with 4 passes (Active Comparator): biopsy with 4 passes of the needle
  Interventions: Procedure: EUS FNA with 4 passes

INTERVENTIONS:
Procedure: EUS FNA with 2 passes — biopsy with 2 passes
  Other Names: Biopsy; FNA
  Arms: EUS FNA with 2 passes
Procedure: EUS FNA with 4 passes — biopsy with 4 passes
  Other Names: biopsy; FNA
  Arms: EUS FNA with 4 passes

SUMMARY:
This study will test the amount of tissue, called "cell block", obtained from your pancreas. Patients who are asked to participate in this study have a growth (mass) in the pancreas that needs a biopsy so a diagnosis can be made. Although we usually perform 2 to 4 passes (number of times the doctor biopsies the mass), at this time we do not know the ideal number of passes needed to obtain adequate amount of tissue for making a diagnosis. The purpose of this study is to compare the amount of tissue obtained with 2 passes versus 4 passes.

DETAILED DESCRIPTION:
Primary Aim:

To compare the number of passes required for obtaining adequate cell block material during EUS-guided FNA of solid pancreatic mass lesions.

Primary Research Hypothesis:

More specimen is required to obtain definitive diagnosis on cell block. This translates to less need for repeat procedures (due to nondiagnostic index procedure due to inadequate FNA passes), prompt treatment to patients and better use of health care resources. Therefore, we will be comparing 2 versus 4 FNA passes to determine which number of FNA pases will yield an adequate diagnostic cell block.

Secondary Aims:

To compare the rate of complications when performing 2 versus 4 EUS-FNA passes of solid pancreatic mass lesions.

Secondary Research Hypothesis:

EUS-guided FNA is a safe procedure with a complication rate of < 1%. By performing more (four) NA passes one is likely to yield a better quality cell block while at the same time without compromising patient safety.

ELIGIBILITY:
Inclusion Criteria:

1) All patients referred to Florida Hospital Endoscopy Unit for assessment of pancreatic mass lesions that require FNA.

Exclusion Criteria:

1. Age <19 years
2. Unable to safely undergo EUS for any reason
3. Coagulopathy (INR >1.6, Prothrombin Time >18secs, Thrombocytopenia <80,000 cells/ml)
4. Unable to consent
5. Non-English speaking patients.
6. Participation in any other Clinical Trial (excluding registries and databases)

Ages: 19 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
number of passes | up to 12 months
  The primary endpoint of the study is to compare the number of passes required to make definitive diagnosis on cell block. This will be assessed by amount (quantity) of the sample to make the diagnosis proportionate to which group the subject was randomized to (two passes versus four passes).

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth
Locations (1):
- Florida Hospital, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varadarajulu S, Bang JY, Holt BA, Hasan MK, Logue A, Hawes RH, Hebert-Magee S. The 25-gauge EUS-FNA needle: Good for on-site but poor for off-site evaluation? Results of a randomized trial. Gastrointest Endosc. 2014 Dec;80(6):1056-63. doi: 10.1016/j.gie.2014.05.304. Epub 2014 Jun 25. PMID 24973173